CLINICAL TRIAL: NCT00932425
Title: Long-term Cardiac Monitoring After Cryptogenic Stroke (CMACS): A Pilot Randomized Trial
Brief Title: Long-term Cardiac Monitoring After Cryptogenic Stroke (CMACS)
Acronym: CMACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CMACS
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Stroke
Keywords: Stroke; Cryptogenic; Cardioembolic; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient cardiac monitoring (Experimental): Patients will be assigned to wear a portable outpatient cardiac telemetry device for 21 days
  Interventions: Device: Cardionet Mobile Cardiac Outpatient Telemetry (MCOT)
- Control (No Intervention): Patients will be discharged home with standard clinical follow-up

INTERVENTIONS:
Device: Cardionet Mobile Cardiac Outpatient Telemetry (MCOT) — Patients will be assigned to wear the telemetry device for 21 days
  Arms: Outpatient cardiac monitoring

SUMMARY:
Atrial fibrillation (AF) is a common and treatable cause of ischemic stroke, but it can be paroxysmal and asymptomatic, and therefore difficult to detect. Patients with stroke routinely undergo 24 hours of continuous cardiac telemetry during hospitalization for stroke as a means of excluding AF. Small studies indicate that extending the duration of monitoring with portable outpatient telemetry devices detects more cases of AF. However, these studies are small and lack control groups, and cannot demonstrate that prolonged cardiac monitoring detects more cases of AF than routine clinical follow-up. The investigators therefore propose a pilot study to determine the feasibility of randomizing patients to prolonged cardiac monitoring or routine clinical follow-up. The investigators will enroll 40 consecutive adult patients seen at the University of California at San Francisco (UCSF) Neurovascular service with cryptogenic stroke or high-risk TIA (ABCD2 score 4 or greater). Enrolled patients will be randomized in a 1:1 fashion. Group A will be assigned to wear an ambulatory cardiac event monitor for 21 days. Group B will be discharged home without a monitor and will serve as controls during routine clinical follow-up. The investigators' primary outcome will be feasibility, defined as more than 80% of randomized patients completing full clinical follow-up and more than 70% of cardiac monitoring if applicable. The investigators' secondary outcomes will be diagnoses of AF at 90 days and 1 year and diagnoses of recurrent stroke at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Seen at UCSF Medical Center for cryptogenic stroke or high-risk TIA
* Onset of stroke or TIA symptoms within the previous 60 days

Exclusion Criteria:

* Definite small-vessel etiology by history or imaging
* Source found on vascular imaging of possible culprit vessels
* Source found by echocardiography (TEE not required)
* History of atrial fibrillation
* Atrial fibrillation on admission ECG
* Atrial fibrillation detected by inpatient cardiac telemetry (at least 24 hours required)
* Obvious culpable systemic illness such as endocarditis
* Patient unable to provide written, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wade Smith, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 patients were enrolled between October 29, 2009 and May 24, 2011
Groups:
- Outpatient Cardiac Monitoring: Patients assigned to wear a portable outpatient cardiac telemetry device for 21 days
  Cardionet Mobile Cardiac Outpatient Telemetry (MCOT): Patients will be assigned to wear the telemetry device for 21 days
- Control: Patients discharged home with standard clinical follow-up
Period: Overall Study
Arm/Group | Outpatient Cardiac Monitoring | Control
Started | 20 | 20
Completed | 20 | 18
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: per protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Outpatient Cardiac Monitoring | Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (15) | 69 (9) | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Completion of Clinical Follow-up as a Measure of Feasibility
Description: Feasibility was defined as 90% or more of randomized patients completing full clinical follow-up and 70% or more completion of assigned cardiac monitoring if applicable
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Outpatient Cardiac Monitoring | Control
Number analyzed (Participants) | 20 | 20
participants | 20 | 18

2. Secondary Outcome: Diagnosis of Atrial Fibrillation
Time Frame: 90 days
Population: 2 patients in the control arm did not have a full 90 days of assessment (see Participant Flow)
Measure: Number; unit: participants
Arm/Group | Outpatient Cardiac Monitoring | Control
Number analyzed (Participants) | 20 | 18
participants | 0 | 0

3. Secondary Outcome: Diagnosis of Atrial Fibrillation
Time Frame: 1 year
Population: 2 participants in the Control arm were followed for less than 90 days
Measure: Number; unit: participants
Arm/Group | Outpatient Cardiac Monitoring | Control
Number analyzed (Participants) | 20 | 18
participants | 0 | 0

4. Secondary Outcome: Recurrent Stroke or TIA
Description: Patients and their primary physicians or neurologists were contacted at 3 months and 1 year after discharge and reported clinical diagnoses of recurrent stroke or TIA using validated questionnaires. Reported events were verified by review of relevant medical records.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Outpatient Cardiac Monitoring | Control
Number analyzed (Participants) | 20 | 18
participants
  Stroke | 0 | 1
  TIA | 1 | 2

5. Primary Outcome: Completion of Assigned Monitoring as a Measure of Feasibility
Description: Feasibility criteria included more than 70% completion of cardiac monitoring if applicable. Patients in the Monitoring arm were assigned to wear a Cardionet mobile cardiac outpatient telemetry monitor for 21 days. Outpatient monitoring began 22 days (+/- 12 days) after symptom onset.
Time Frame: 21 days
Population: Only patients in the monitoring arm were assessed for compliance with assigned monitoring
Measure: Number; unit: participants
Arm/Group | Outpatient Cardiac Monitoring
Number analyzed (Participants) | 20
participants | 15

ADVERSE EVENTS:
Time Frame: 1 year
Description: Participants were assessed for adverse events attributable to the intervention during the monitoring period, and for recurrent stroke or TIA at 3 months and 1 year
Arm/Group | Outpatient Cardiac Monitoring | Control
Serious Adverse Events (participants affected / at risk) | 1/20 | 3/18
Other Adverse Events (participants affected / at risk) | 1/20 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatient Cardiac Monitoring (N=20) | Control (N=18)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
TIA (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatient Cardiac Monitoring (N=20) | Control (N=0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One participant in the monitoring group had contact dermatitis, which we classified as an AE attributable to the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No